CLINICAL TRIAL: NCT00368875
Title: Phase I/II Study of a Combination of Suberoylanilide Hydroxamic Acid (Vorinostat) Plus Paclitaxel and Bevacizumab in Patients With Advanced Metastatic and/or Local Chest Wall Recurrent Breast Cancer
Brief Title: Phase I-II Study of Vorinostat, Paclitaxel, and Bevacizumab in Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03012; NCI-2012-03012 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 06-05-291 (Other: Montefiore Medical Center); 7703 (Other: CTEP); N01CM62204 (NIH); N01CM62207 (NIH); N01CM62205 (NIH); N01CM62209 (NIH)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2014-03

CONDITIONS: Male Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Vorinostat; Paclitaxel; Taxes; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vorinostat, paclitaxel, bevacizumab (Experimental): Vorinostat BID on days 1-3, 8-10, and 15-17, paclitaxel IV over 1 hour on days 2, 9, and 16, bevacizumab IV over 30-90 minutes on days 2 and 16, repeat every 28 days.
  Interventions: Drug: vorinostat; Drug: paclitaxel; Biological: bevacizumab

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF

SUMMARY:
This phase I/II trial is studying the side effects and best dose of vorinostat when given together with paclitaxel and bevacizumab and to see how well they work in treating patients with metastatic breast cancer and/or breast cancer that has recurred in the chest wall and cannot be removed by surgery. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving vorinostat together with paclitaxel and bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRiMARY OBJECTIVES:

I. To determine the recommended phase II dose of oral suberoylanilide hydroxamic acid (vorinostat) in combination with weekly paclitaxel and bevacizumab in patients with chest wall recurrent or metastatic breast cancer. (Phase I) II. To determine the efficacy (response rate, response duration, time to disease progression, time to treatment failure, and overall survival) and toxicity of oral suberoylanilide hydroxamic acid (vorinostat) in combination with weekly paclitaxel and bevacizumab in patients with chest wall recurrent or metastatic breast cancer. (Phase II)

SECONDARY OBJECTIVES:

I. To determine whether in vivo treatment with vorinostat induces a) acetylation of proteins including histone H3 and H4, b) ubiquitylation of proteins, and c) the levels of p21 and p27 levels in the peripheral blood mononuclear cells (pre treatment vs. cycle 1 day 2 after 3 VORINOSTAT doses but prior to paclitaxel.

II. To determine whether in vivo treatment with vorinostat induces a) acetylation of proteins including histone H3 and H4, ubiquitylation of proteins, and c) the levels of Bim, Bak, tBID, p21 and p27 levels, as well as down regulate Bcl-2, Bcl-xL and survivin in chest wall recurrent or metastatic breast cancer cells (pre treatment vs. cycle 1 day 2 after 3 vorinostat doses but prior to paclitaxel).

III. To determine whether in the primary breast cancer (and metastatic cancer if available) pretreatment levels of Her-2, Estrogen Receptor (ER)-alpha, Progesterone Receptor (PR), p21, p27, p-AKT, p-ERK1/2, HDAC1, 2, 3, 4, 6, 10 and SIRT2 levels predict for the response to treatment with VORINOSTAT plus paclitaxel.

OUTLINE: This is a phase I, multicenter, dose-escalation study of vorinostat (SAHA) followed by a phase II, open-label study.

Phase I: Patients receive oral SAHA twice daily on days 1-3, 8-10, and 15-17, paclitaxel IV over 1 hour on days 2, 9, and 16, and bevacizumab IV over 30-90 minutes on days 2 and 16. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. The recommended phase II dose is defined as one dose level below the MTD.

Phase II: Patients receive SAHA at the recommended phase II dose and paclitaxel and bevacizumab as in phase I.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed adenocarcinoma of the breast; effective with version 2.2 (1/26/09), only patients with disease that is accessible to biopsy and consent to serial biopsy are eligible
* stage IV disease, locally recurrent inoperable chest wall disease; at least one bidimensional and/or unidimensional, measurable indicator lesion must be present (patients with only non-measurable disease are eligible for the phase I trial only); all sites of disease should be noted and followed
* ECOG performance status =< 1 (Karnofsky >= 70%)
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 100,000/ul
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 x institutional upper limit of normal
* PTT and either INR or PT < 1.5 x normal
* Creatinine within normal institutional limits OR creatinine clearance >= mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Urine protein should be screened by urine analysis for Urine Protein Creatinine (UPC) ratio; for UPC ratio > 0.5, 24-hour urine protein should be obtained and the level should be < 1000 mg for patient enrollment;
* LVEF must be at or above the lower institutional limit of the normal range (on MUGA or Echo obtained within 12 weeks of registration, or within 4 weeks of prior Herceptin)
* Not pregnant/lactating

Exclusion criteria:

* chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* may not be receiving any other investigational agents.
* history of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat or other agents used in the study (e.g., paclitaxel, bevacizumab, quinolones)
* uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sparano, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Result] Ramaswamy B, Fiskus W, Cohen B, Pellegrino C, Hershman DL, Chuang E, Luu T, Somlo G, Goetz M, Swaby R, Shapiro CL, Stearns V, Christos P, Espinoza-Delgado I, Bhalla K, Sparano JA. Phase I-II study of vorinostat plus paclitaxel and bevacizumab in metastatic breast cancer: evidence for vorinostat-induced tubulin acetylation and Hsp90 inhibition in vivo. Breast Cancer Res Treat. 2012 Apr;132(3):1063-72. doi: 10.1007/s10549-011-1928-x. Epub 2011 Dec 27. PMID 22200869

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July 2006 and December 2009 a total of 54 patients were registered on the study.
Groups:
- Phase I: Vorinostat dose (200 or 300 mg BID) was assigned at the time of registration. Vorinostat was administered orally twice daily on days 1-3, 8-10, and 15-17 of each 28-day cycle.
  All patients also received paclitaxel at 90 mg/m2 as 1-hour infusion on days 2, 9, and 16 of every 28-day cycle. Bevacizumab was administered on day 2 and day 16 of the 28 day cycle at 10 mg/kg dose. Vorinostat dose escalation was carried out in the standard 3 + 3 phase I trial design based upon toxicity observed during the first cycle of therapy.
- Phase II: Vorinostat was administered orally twice daily at the recommended phase II dose of 300 mg on days 1-3, 8-10, and 15-17 of each 28-day cycle.
  All patients also received paclitaxel at 90 mg/m2 as 1-hour infusion on days 2, 9, and 16 of every 28-day cycle. Bevacizumab was administered on day 2 and day 16 of the 28 day cycle at 10 mg/kg dose.
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 6 | 48
Completed | 0 | 0
Not Completed | 6 | 48
Not completed — Adverse Event | 0 | 12
Not completed — Progressive disease | 3 | 27
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Other Reason | 0 | 2
Not completed — Alternative Therapy | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I + Phase II: Phase I: Vorinostat dose (200 or 300 mg BID) was assigned at the time of registration. Vorinostat was administered orally twice daily on days 1-3, 8-10, and 15-17 of each 28-day cycle.
  All patients also received paclitaxel at 90 mg/m2 as 1-hour infusion on days 2, 9, and 16 of every 28-day cycle. Bevacizumab was administered on day 2 and day 16 of the 28 day cycle at 10 mg/kg dose. Vorinostat dose escalation was carried out in the standard 3 + 3 phase I trial design based upon toxicity observed during the first cycle of therapy.
  Phase II: Vorinostat was administered orally twice daily at the recommended phase II dose of 300 mg on days 1-3, 8-10, and 15-17 of each 28-day cycle.
  All patients also received paclitaxel at 90 mg/m2 as 1-hour infusion on days 2, 9, and 16 of every 28-day cycle. Bevacizumab was administered on day 2 and day 16 of the 28 day cycle at 10 mg/kg dose.
Arm/Group | Phase I + Phase II
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 54 [27 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 37
  Black | 11
  Asian | 2
  Unknown | 4

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose as Assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 (Phase I)
Description: Dose-limiting toxcities (DLT) were defined as grade 3-4 febrile neutropenia, thrombocytopenia and non-hemtological toxicity attributed to therapy (nausea, vomiting and diarrhea would be considered dose limiting only if not adequately controlled with therapy). Any toxicity occurring during cycle 1 that resulted in dose reduction of vorinostat or paclitaxel or failure to complete all protocol specificed doses in the first cycle was also considered a DLT
Time Frame: 28 days
Population: Three patients were treated at the first vorinostat dose level of 200 mg BID and three additional patients were treated at the second dose level of 300 mg BID
Measure: Number; unit: mg
Arm/Group | Phase I
Number analyzed (Participants) | 6
mg | 300

2. Primary Outcome: Objective Response Rate (CR + PR)
Description: Estimated and a 95% confidence interval will be estimated via binomial proportions. Per Response Evaluation Criteria in Solid Tumors (RECIST) for target lesions and assessed by CT scan: Complete response (CR): Disappearance of all target lesions; Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR+PR.
Time Frame: Up to 12 months
Population: 53 patients in the phase I and phase II portions were evaluated. One patient was not eligible to be evaluated for objective response rate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I + Phase II
Number analyzed (Participants) | 53
percentage of participants | 49 [37 to 60]

3. Secondary Outcome: Progression-free Survival (PFS),
Description: Assessed by Kaplan-Meier survival analysis and 95% confidence intervals will be calculated using Greenwood's formulae.
Time Frame: From first treatment day until objective or symptomatic progression, assessed up to 12 months
Population: 53 patients in the phase I and phase II portions were evaluated
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I + Phase II
Number analyzed (Participants) | 53
months | 11.9 [8.9 to 13.9]

4. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Assessed by Kaplan-Meier survival analysis and 95% confidence intervals will be calculated using Greenwood's formulae. Time to treatment failure was not reported for this study.
Time Frame: Time from the first treatment day until disease progression or discontinuation of treatment due to toxicity, assessed up to 12 months
Population: Zero participants analyzed because time to treatment failure was not assessed.
Arm/Group | Vorinostat, Paclitaxel, Bevacizumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival(OS)
Description: Assessed by Kaplan-Meier survival analysis and 95% confidence intervals will be calculated using Greenwood's formulae.
Time Frame: Time from first treatment day until death, assessed up to 12 months
Population: 54 patients in the phase I and phase II portion were evaluated
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I
Number analyzed (Participants) | 54
months | 29.4 [25.6 to 34.7]

ADVERSE EVENTS:
Arm/Group | Phase I + Phase II
Serious Adverse Events (participants affected / at risk) | 27/54
Other Adverse Events (participants affected / at risk) | 40/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I + Phase II (N=54)
Neutropenia (Blood and lymphatic system disorders) | 15
Anemia (Blood and lymphatic system disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Headache (General disorders) | 3
Fatigue (General disorders) | 10
Neuropathy (Nervous system disorders) | 12
Proteinuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I + Phase II (N=54)
Anemia (Blood and lymphatic system disorders) | 20
Neutropenia (Blood and lymphatic system disorders) | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Vomiting (Gastrointestinal disorders) | 21
Diarrhea (Gastrointestinal disorders) | 40
Fatigue (General disorders) | 35
Neuropathy (Nervous system disorders) | 25
Epistaxis (Ear and labyrinth disorders) | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less